CLINICAL TRIAL: NCT01535651
Title: Using Social Media to Enhance the Impact of the Teen Outreach Program
Acronym: TOP4ME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado School of Public Health (Other)
Collaborators: Denver Health and Hospital Authority (Other)
Responsible Party: Principal Investigator, Sheana Bull, Professor, Colorado School of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OAH Denver Health
Record Dates: First submitted 2012-02-15; First posted 2012-02-20 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Pregnancy Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TOP Program plus Text messaging (Experimental): Boys and Girls Club members who participate in TOP over 9 months will receive regular text messages in addition to TOP
  Interventions: Behavioral: Teen Outreach Program with Media Enhancement (TOP4ME)
- TOP Program alone (No Intervention): Boys and Girls Club participants will participate in TOP for 9 months

INTERVENTIONS:
Behavioral: Teen Outreach Program with Media Enhancement (TOP4ME) — Persons participating in TOP will receive text messages weekly in addition to TOP
  Other Names: Youth All Engaged! (YAE!)
  Arms: TOP Program plus Text messaging

SUMMARY:
The investigators are exploring the use of short message service (text) messaging by cell phones to enhance the effects of the Teen Outreach Program, an effective teen pregnancy prevention program.

ELIGIBILITY:
Inclusion Criteria:

* boys and girls club member in metro Denver, age 14-18

Exclusion Criteria:

* non-english speaking

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 852 (Actual)
Dates: Start 2011-09; Primary Completion 2015-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
pregnancy | 21 months

SECONDARY OUTCOMES:
school drop out | 21 months

CONTACTS AND LOCATIONS:
Locations (1):
- Boys and Girls Clubs of Metro Denver, Denver, Colorado, United States

REFERENCES:
- [Background] Devine S, Bull S, Dreisbach S, Shlay J. Enhancing a Teen Pregnancy Prevention Program with text messaging: engaging minority youth to develop TOP (R) Plus Text. J Adolesc Health. 2014 Mar;54(3 Suppl):S78-83. doi: 10.1016/j.jadohealth.2013.12.005. PMID 24560081